CLINICAL TRIAL: NCT05278611
Title: A Randomized, Double-blind, Placebo-controlled Dose Escalation Phase Ia Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of EP-9001A Injection in Healthy Subjects
Brief Title: a Safety and Tolerability Study of EP-9001A in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Easton Biopharmaceuticals Co,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EP-9001A-Ia
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP-9001A (Experimental): Dose-escalation trial
  Interventions: Drug: EP-9001A
- Placebo (Placebo Comparator): Dose-escalation trial
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EP-9001A — The initial dose of the study was set as 1 mg, and the doses were escalated sequentially in the order of 1 mg, 2.5 mg, 5 mg, 10 mg, 20 mg, and 25 mg
  Other Names: NGF mab
  Arms: EP-9001A
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
Nerve Growth Factor（NGF）plays an important role in the pathogenesis of neuropathic pain including cancer pain. EP-9001A is a humanized monoclonal antibody targeting NGF, thus thought to alleviate neuropathic pain though the blockade of NGF signal pathway.

The primary objective of the study is to assess the safety and tolerability of a single dose of subcutaneous (SC) administered EP-9001A in healthy Chinese subjects.

DETAILED DESCRIPTION:
Nerve Growth Factor（NGF）plays an important role in the pathogenesis of neuropathic pain including cancer pain. EP-9001A is a humanized monoclonal antibody targeting NGF, thus thought to alleviate neuropathic pain though the blockade of NGF signal pathway.

The primary objective of the study is to assess the safety and tolerability of a single dose of subcutaneous (SC) administered EP-9001A in healthy Chinese subjects.

The initial dose of the study was set as 1 mg, and the doses were escalated sequentially in the order of 1 mg, 2.5 mg, 5 mg, 10 mg, 20 mg, and 25 mg

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female Chinese volunteers ≥18 and ≤45 years of age at the screening visit;
2. Body weight ≥ 45.0 kg for female subjects and ≥ 50.0 kg for male subjects with a body mass index (BMI) between 19.0 and 26.0 kg/m2( including border value);
3. Subjects during the trial (female subjects from 14 days before dosing, male subjects from dosing) to 3 months after the end of the trial without fertility or sperm/egg donation plan and voluntarily take effective physical contraception measures;
4. According to the results of physical examination, vital signs, ECG and clinical laboratory tests during the screening period, all the test results are normal or abnormal without clinical significance as judged by the investigator;
5. Signed a written informed consent.

Exclusion Criteria:

1. history of allergic diseases (including but not limited to asthma, urticaria, allergic rhinitis), or a history of drug allergy, or a history of allergy to the test drug ingredients;
2. history of clinical serious diseases and not cured, such as motor (muscle and bone) system, digestive system, respiratory system, genitourinary system, blood (hematopoietic) system, circulatory system, nervous system, mental system, endocrine system, cardiovascular system and metabolic abnormalities;
3. received surgery in the past 3 months or have surgery plan during the trial ;
4. Have used any prescription, over-the-counter or health care products in the past 2 weeks;
5. took more than 10 cigarettes a day or the same amount of tobacco or can not stop tobacco during trial;
6. alcohol breath test positive;
7. History of alcohol abuse within the past 6 months;
8. History of drug abuse, positive results of urine multiple drug tests;
9. Drink excessive tea, grapefruit juice, coffee or caffeinated beverages (an average of more than 8 cups per day, 200 mL per cup) every day in the past 1 month;
10. Participated in other drug clinical trials in the past 3 months, or plan to participate in other clinical trials during this study;
11. Blood loss/blood donation of more than 400 mL in the past 3 months (except for female physiological blood loss), or receiving blood transfusion or use of blood products, or planning to donate blood during the trial or within 1 month after the end of the trial;
12. Vaccinated within the past 1 month
13. positive in Hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus antibody, syphilis specific antibody screening;
14. Subjects who are lactating, pregnant or plan to become pregnant or conceive recently;
15. Patients with a history of bone or joint diseases, including but not limited to osteoarthritis, pathological fractures, osteonecrosis, rheumatoid arthritis, neuropathic arthritis, lupus erythematosus or inflammatory joint diseases;
16. Patients with a history of joint-related events, such as total joint replacement (TJR) surgery, meniscus or knee ligament injury (with or without surgical repair) or joint infection, or bone dislocation, hip dislocation, knee dislocation within 1 year before screening;
17. Kellgren-Lawrence grade ≥ 2 in any major joint (shoulder, hip, knee);
18. History of clinically significant peripheral neuropathy, paresthesia, dysesthesia;
19. History of autonomic neuropathy or diabetic neuropathy;
20. The investigator assesses the poor compliance, or the investigator believes that the subject has any other conditions that are not suitable for participating in this clinical study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number and severity of Adverse Events，MTD | Baseline to week 8
  All adverse events occurring throughout the study were assessed and graded. the maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
pharmacokinetics of EP-9001A | Baseline to week 8
  EP-9001A serum concentrations over time
immunogenicity assessed by ADA | Baseline to week 8
  Presence of anti-drug antibodies over time

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No